CLINICAL TRIAL: NCT05971264
Title: Comparison of Bladder Pressure Versus Regional Intestinal Tissue Oxygenation in Infants
Acronym: BPvsNIRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1002
Record Dates: First submitted 2023-05-15; First posted 2023-08-02 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Intraabdominal Hypertension; Abdominal Compartment Syndrome
Keywords: Near infra-red spectroscopy; Bladder pressure; Intraabdominal pressure
MeSH Terms: conditions — Intra-Abdominal Hypertension | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Diagnostic Test: Near infrared-spectroscopy

INTERVENTIONS:
Diagnostic Test: Near infrared-spectroscopy — Comparison of regional intestinal oxygen saturation (measured with near infrared-spectroscopy) and indirect intraabdominal pressure measurement (bladder pressure) in muscle-relaxed, sedated patients compared to awake, non-sedated patients.

SUMMARY:
The goal of this clinical trial is to learn more about intestinal regional oxygen saturation measurements made with near-infrared spectroscopy and bladder pressure measurements in infants without risk of intraabdominal hypertension. The main question it aims to answer is if - in comparison to bladder pressure - the regional intestinal oxygen saturation measured with near-infrared spectroscopy is stable in the muscle-relaxed, intubated patients and the awake and non-sedated patient.

In case of participation the bladder pressure and the regional intestinal oxygen saturation (measured with near-infrared spectroscopy) will each be measured once intraoperatively and once postoperatively. Patients included in this study will be undergoing an operation which necessitates muscle-relaxation, as well as an indwelling urinary catheter during the operation and for a short-time thereafter for other reasons than this study.

ELIGIBILITY:
Inclusion Criteria:

* Prepped and consented for laparoscopic pyeloplasty or minimal PSARP with perineal or vestibular fistula or lateral thoracotomy for the correction of esophageal atresia
* Age of 12 months old or less at operation
* Legal custodian gives consent

Exclusion Criteria:

* Anterior abdominal wall thickness greater than 12 mm measured on preoperative MRI imaging if available
* Patients planned for additional intestinal surgeries or non-standard pyeloplasty, e.g. pyeloplasty with nephrostoma
* Patients planned for laparoscopic pyeloplasty whose intraoperative urine sample shows pathological results
* Patients with esophageal atresia who experience pulmonary decompensation and need urgent surgery for fistula clipping

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intestinal rSpO2 measurements in muscle-relaxed, intubated patients | intraoperative measurements taken within the first 10 minutes after anaesthesia induction
  Our primary endpoint is the regional intestinal oxygen saturation (rSpO2) measurement (average of 5 measurements taken every 30 seconds within 2 minutes) in muscle-relaxed, intubated patients
Intestinal rSpO2 measurements in awake, non-sedated patients | postoperative measurements taken within the first three postoperative days
  Our primary endpoint is the regional intestinal oxygen saturation (rSpO2) measurements (average of 5 measurements taken every 30 seconds within 2 minutes) in awake, non-sedated patients

SECONDARY OUTCOMES:
Bladder pressure values | taken once intraoperatively within the first 10 minutes after anaesthesia induction and once postoperatively within the first three postoperative days
  Bladder pressure measurements measured under two different circumstances: once muscle-relaxed, intubated patients (i.e. under ideal circumstances for these measurements) and once in awake, non-sedated patients (less ideal circumstances).

CONTACTS AND LOCATIONS:
Overall Officials: Hannah R Neeser, MD, Principal Investigator — University Children's Hospital of Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No